CLINICAL TRIAL: NCT01949506
Title: Pilot Study Evaluating Stereotactic Body Radiation Therapy (SBRT) and Adaptive Radiation Therapy (ART) for Pulmonary Metastases From Soft Tissue Sarcomas
Brief Title: (SBRT) and (ART) for Pulmonary Metastases From Soft Tissue Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Meena Bedi, Principal Investigator, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00020337
Record Dates: First submitted 2013-09-04; First posted 2013-09-24 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Stage IV Adult Soft Tissue Sarcoma; Sarcoma,Soft Tissue
Keywords: Lung metastases; Radiation Therapy; Stereotactic Body Radiation Therapy; Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Body Radiation Therapy (Other): Arms: Stereotactic Body Radiation Therapy (SBRT) with Adaptive Radiation Therapy (ART) for all patients. A non-randomized study. Patients must have 1-5 pulmonary metastases all less than 5 cm in size. Pathologic confirmation of primary soft tissue sarcoma. All lesions to receive 3-5 fractions to each tumor. Treatments delivered with > 10 Gy per fraction will have a minimum of 48 hour interfraction interval. For treatments with ≤ 10 Gy per fraction will have a minimum 24 hour interfraction interval. Treatments will be ideally completed over 14 days for 3 fraction treatments and over 21 days for >5 fraction treatment schedules.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
This is a prospective study to document the local control rates with SBRT specifically for pulmonary metastases from soft tissue sarcoma. This study will prospectively document acute and late toxicity, quality of life (QoL), tumor control, and survival.

DETAILED DESCRIPTION:
A total of no more than 20 people are expected to participate in this study at the Medical College of Wisconsin/Froedtert Hospital. Patients will be followed for three years.

The usual treatment for sarcomas that spread to the lungs is to remove the cancer with surgery. Patients who cannot have surgery or prefer not to have surgery, can receive radiation therapy. Standard radiation therapy involves several weeks of daily treatment sessions, although it is not as effective as surgery and may seriously damage normal surrounding lung tissue. Stereotactic body radiation therapy (SBRT) is a radiation treatment that gives fewer but higher doses of radiation than standard radiation. SBRT is used to treat metastases to the lung from many types of cancer but has not been used very often with patients who have metastatic disease to their lungs from sarcomas.

The purpose of this study is to test the possibility of SBRT to the lung for metastatic disease to the lung. This information will be used to find out if there are factors that can predict recovery or outcome of patients with metastatic disease to the lung from sarcoma. SBRT will consist of 1 to 3 treatments per week for a total of 3 to 5 treatments to each tumor until therapy is complete. After SBRT is completed, follow-up exams will occur 4-6 weeks from the completion of radiation treatment, every 3 months in year 1 and every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Pathologic confirmation of primary soft tissue sarcoma with pathologic or radiographic evidence of pulmonary metastatic disease
* No evidence of extra pulmonary progression of disease for 3 months prior to enrollment on study
* 1-5 pulmonary lesions all ≤5 cm in size
* Medically inoperable or declines surgery
* Patients may have had previous treatment for pulmonary metastases

Exclusion Criteria:

* Patients who have uncontrolled extra-pulmonary disease
* Pregnant women
* Patients who have greater than 5 pulmonary lesions at the time of study enrollment
* Patients who have disease progression outside the lungs within 3 months of enrollment on the study
* Disease pathology other than sarcoma subtypes
* Patients with a history of metastatic disease from a primary other than sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Bedi, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy
Started | 9
Completed | 8
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events of Grade ≥ 3 by CTCAE Criteria.
Description: This measure (number of adverse events of grade ≥ 3 by Common Terminology Criteria for Adverse Events (CTCAE) criteria) will provide information regarding the acute toxicity of SBRT for < 5 pulmonary metastases from soft tissue sarcoma..The CTCAE criteria provide a standardized description of adverse events including guidelines for grading severity. The guidelines can be viewed at: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm.
Time Frame: 6 weeks post SBRT
Measure: Number; unit: events
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 8
events | 8

2. Secondary Outcome: Number of Subjects Experiencing Locoregional Recurrences.
Description: This measure (number of subjects experiencing locoregional recurrences) will provide information regarding locoregional control. Locoregional recurrence means any new or renewed tumor growth of any size observed by an imaging technology that is located at or adjacent to a prior treatment site.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 8
Participants | 0

3. Other Pre Specified Outcome: Quality of Life Questionnaire Score
Description: Quality of life will be measured using the Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire. The FACT-L is a statistically validated, 36-question, Likert-type instrument using a five-point scale from 0 (not at all) to 4 (very much). The questionnaire assesses 5 domains: physical, social/family, emotional, and functional well-being; and lung cancer subscale (symptoms, cognitive function, regret of smoking). The subscale scores are added to determine the total score. The scoring range is 0-28 with higher numbers indicating more severe outcomes.
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months, and 36 months
Population: Of the 8 subjects in the study, 3 expired within the 3-year timeframe. At their 36-month visit, 2 additional subjects did not complete the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 8
units on a scale
  Baseline | 17.1 (1.5)
  6 Months: number analyzed (Participants) | 6
  6 Months | 16.7 (3.2)
  12 Months: number analyzed (Participants) | 5
  12 Months | 16.3 (1.9)
  18 Months: number analyzed (Participants) | 5
  18 Months | 16.4 (1.5)
  24 Months: number analyzed (Participants) | 5
  24 Months | 17.0 (1.5)
  36 Months: number analyzed (Participants) | 3
  36 Months | 17.1 (1.1)

4. Other Pre Specified Outcome: Overall Survival
Description: This measure is the number of subjects alive at three years.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 8
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (N=8)
Disease progression (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Body Radiation Therapy (N=8)
Anxiety (Psychiatric disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Burning sensation in chest (General disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT01949506/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT01949506/ICF_001.pdf